CLINICAL TRIAL: NCT00832000
Title: Phase II Therapeutic Trial of Mexiletine in Non-Dystrophic Myotonia
Brief Title: Effectiveness of Mexiletine for Treating People With Non-Dystrophic Myotonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Richard Barohn, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Barohn, MD, Gertrude and Dewey Zeigler Professor of Neurology and Chair, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11050; FDA OPD RO1FD003454; NCT00721942 (obsolete NCT alias)
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Myotonia; Non-Dystrophic Myotonia
MeSH Terms: conditions — Myotonia | interventions — Mexiletine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive mexiletine for 4 weeks, then no intervention for 1 week, and finally placebo for 4 weeks.
  Interventions: Drug: Mexiletine; Drug: Placebo
- 2 (Experimental): Participants will receive placebo for 4 weeks, then no intervention for 1 week, and finally mexiletine for 4 weeks.
  Interventions: Drug: Mexiletine; Drug: Placebo

INTERVENTIONS:
Drug: Mexiletine — 200 mg three times a day; in pill form
Drug: Placebo — Placebo three times a day; in pill form

SUMMARY:
Nondystrophic myotonias (NDM) are neuromuscular disorders caused by genetic abnormalities in certain muscle cell membrane proteins. The proteins affect muscle contraction. Individuals with NDM experience limited muscle relaxation, which then can cause pain, weakness, incoordination, and impaired physical activity and function. Because NDM is very rare, information on the best way to treat people with the disorders is lacking, and there are no FDA-approved therapies. The purpose of this study is to determine the effectiveness of the medication mexiletine in treating people with NDM.

DETAILED DESCRIPTION:
NDM are neuromuscular disorders that are caused by mutations in skeletal muscle ion channels, usually voltage-dependent sodium and chloride channels. The poorly functioning channels result in impaired muscle relaxation after contraction, which is also called myotonia. Mexiletine is an antiarrhythmic medication that has a high affinity for muscle sodium channels and may have the ability to correct delayed inactivation of sodium channels. In case reports and single-blind clinical trials, mexiletine was shown to reduce symptoms of myotonia. Currently, there is no standard strategy for treating people with NDM, and effective treatment options are needed. This study will determine the effectiveness of mexiletine in treating people with NDM.

Participation in this study will last 9 weeks and will involve two separate 4-week treatment periods, with a 1-week washout period between them. During the first treatment period, participants will be randomly assigned to receive either mexiletine or placebo, both of which will be taken three times a day. This will be followed by 1 week of no treatment. During the second treatment period, participants will receive whichever treatment they did not receive initially and will follow the same dosing schedule.

Participants will attend five study visits that will occur at screening and Weeks 0, 4, 5, and 9. Screening will include blood and urine sampling, electrocardiography (EKG), and a medical history. The remaining visits will include a physical examination, a grip test, exercise tests, nerve conduction tests, blood sampling, questionnaires, and electromyography (EMG). EKG will be repeated at Weeks 4, 5, and 9. Throughout the study, participants will phone in daily to report their symptoms. There will be no follow-up visits.

Funded by FDAOPD RO1 0003454.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms or signs suggestive of myotonic disorders
* Presence of myotonic potentials on electromyography (EMG)
* Participant in the Non-Dystrophic Natural History study (RDCRN 5303) or a new patient with confirmed non-dystrophic myotonia

Exclusion Criteria:

* Other neurological condition that might affect the assessment of the study measurements
* Genetic confirmation of DM1 (more than 50 repeats of CTG) or DM2
* Existing cardiac conduction defects, as evidenced on EKG, including but not limited to the following conditions: malignant arrhythmia or cardiac conduction disturbances (e.g., second degree AV block, third degree AV block, or prolonged QT interval)
* Existing permanent pacemaker
* Current use of any of the following antiarrhythmic medications for a cardiac disorder: flecainide acetate, encainide, disopyramide, procainamide, quinidine, propafenone, or mexiletine
* Use of medications for myotonia, such as phenytoin and flecainide acetate, within 5 days of study entry; carbamazepine and mexiletine within 3 days of study entry; or propafenone, procainamide, disopyramide, quinidine, and encainide within 2 days of study entry
* Use of medications that produce myotonia, which may include fibrate acid derivatives, hydroxymethylglutaryl CoA reductase inhibitors, chloroquine, and colchicines
* Kidney or liver disease
* Heart failure
* Seizure disorder
* Pregnant or breastfeeding

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Rochester School of Medicine & Dentistry, Rochester, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- London Health Sciences Center, London, Ontario, Canada
- University of Milan, Milan, Italy
- Institute of Neurology and National Hospital for Neurology, London, United Kingdom

REFERENCES:
- [Derived] Statland JM, Bundy BN, Wang Y, Rayan DR, Trivedi JR, Sansone VA, Salajegheh MK, Venance SL, Ciafaloni E, Matthews E, Meola G, Herbelin L, Griggs RC, Barohn RJ, Hanna MG; Consortium for Clinical Investigation of Neurologic Channelopathies. Mexiletine for symptoms and signs of myotonia in nondystrophic myotonia: a randomized controlled trial. JAMA. 2012 Oct 3;308(13):1357-65. doi: 10.1001/jama.2012.12607. PMID 23032552

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were at least 16 years of age, had clinical symptoms or signs of NDM, and myotonic potentials on electromyography. Participants were either enrolled in the CINCH NDM Natural History Study, or a new patient with genetically confirmed NDM, or with clinical features of NDM but negative myotonic dystrophy DNA testing.
Pre-assignment Details: Patients taking anti-myotonic agents were required to discontinue medications for a wash-out period equal to 7 times the half-life of elimination prior to their baseline visit. Participants were ineligible if they has specific contraindications to taking mexiletine (cardiac conduction defects, hepatic or renal disease, or heart failure).
Groups:
- Mexiletine Then Placebo: 29 Participants will receive mexiletine for 4 weeks, then no intervention for 1 week, and finally placebo for 4 weeks.
  Included in anaysis*: 28 patients
  *Modified intention to treat analysis. 1 subject in each group not included in primary analysis due to failure to make any calls to the IVR system for stiffness in either period
- Placebo Then Mexiletine: 30 Participants will receive placebo for 4 weeks, then no intervention for 1 week, and finally mexiletine for 4 weeks.
  Included in analysis* 29 patients
  *Modified intention to treat analysis. 1 subject in each not included in primary analysis due to failure to make any calls to the IVR system for stiffness in either period.
Period: Overall Study
Arm/Group | Mexiletine Then Placebo | Placebo Then Mexiletine
Started | 29 (Mexiletine 200 mg orally three times daily) | 30 (Placebo)
Crossed Over to Opposite Intervention | 25 (Placebo) | 29 (Mexiletine 200 mg orally three times daily)
Completed | 23 | 29
Not Completed | 6 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No calls to IVR in either period | 1 | 1
Not completed — No calls to IVR in period 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants received all inerventions; therefore, we combined all participants into one Arm/Group.
Arm/Group | All Study Participants
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 56
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 42.9 (25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 31
  Canada | 4
  United Kingdom | 12
  Italy | 12

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Stiffness on the IVR
Description: Stiffness measured on a 1-9 scale, 1 being minimal, 9 the worst ever experienced. 0=no symptom reported. For analysis the average severity of stiffness for each participant was calculated from daily calls made in weeks 3-4 of each period.
Time Frame: Weeks 3-4 of each period
Population: Modified intention to treat analysis (n=57). 2 subjects were excluded from analysis due to failure call the IVR system in either period. Treatment group estimates by period are taken from the mixed model, the number above reflecting the number who contributed to the model point estimate. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mexiletine - Period 1: Mexiletine capsules 200 mg orally three times daily period 1. Due to an interaction between period and treatment the primary outcome was presented separately for periods 1 and 2.
- Placebo - Period 1: Placebo capsules orally three times dailyperiod 1. Due to an interaction between period and treatment the primary outcome was presented separately for periods 1 and 2.
- Mexiletine - Period 2: Mexiletine capsules 200 mg orally three times daily period 2. Due to an interaction between period and treatment the primary outcome was presented separately for periods 1 and 2.
- Placebo - Period 2: Placebo capsules orally three times dailyperiod 2. Due to an interaction between period and treatment the primary outcome was presented separately for periods 1 and 2.
Arm/Group | Mexiletine - Period 1 | Placebo - Period 1 | Mexiletine - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 28 | 29 | 29 | 25
units on a scale | 2.53 [1.80 to 3.17] | 4.21 [3.40 to 5.20] | 1.60 [1.04 to 2.20] | 5.27 [4.44 to 6.27]
Statistical Analysis 1: Comparison: Mexiletine - Period 1 vs Placebo - Period 1; P value indicates significance level of the Wald test associated with mexiletine effect from the linear mixed effects model (n=57). When a carryover effect was detected, the significance level associated with the additive portion of the mexiletine effect (labeled period 1) is followed by the level associated with the interaction of mexiletine and period 2 (labeled period 2). All P values were 2-sided and .05 was considered the threshold of statistical significance; Test type: Superiority or Other; p < 0.001, Wald; Mean Difference (Final Values) = -1.68, 95% CI 2-sided [-2.66 to -0.706], Standard Deviation 1.24 — Residual standard deviation
Statistical Analysis 2: Comparison: Mexiletine - Period 2 vs Placebo - Period 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.04, Wald; Mean Difference (Final Values) = -3.68, 95% CI [-3.85 to -0.139], Standard Deviation 1.24 — Residual standard deviation

2. Secondary Outcome: Patient Reported Pain on the IVR
Description: Pain measured on a 1-9 scale, 1 being minimal, 9 the worst ever experienced. 0=no symptom reported. For analysis the average severity of pain for each participant was calculated from daily calls made in weeks 3-4 of each period.
Time Frame: Weeeks 3-4 of each period
Population: 48 partipants who experienced pain in either period 1 or period 2 were included in analysis. All treatment group means are extracted from the mixed effects model. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mexiletine: Participants experiencing pain on mexiletine capsules 200 mg orally three times daily in period 1 or period 2
- Placebo: Participants experiencing pain on placebo capsules orally three times dailyin period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 48 | 48
units on a scale | 1.54 [0.924 to 2.13] | 3.17 [2.43 to 3.93]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; P value indicates significance level of the Wald test associated with mexiletine effect from the linear mixed effects model. When a carryover effect was detected, the significance level associated with the additive portion of the mexiletine effect (labeled period 1) is followed by the level associated with the interaction of mexiletine and period 2 (labeled period 2). All P values were 2-sided and .05 was considered the threshold of statistical significance; Test type: Superiority or Other; p < 0.001, Wald; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-2.00 to -1.26], Standard Deviation 1.19 — Residual standard deviation

3. Secondary Outcome: Patient Reported Weakness on the IVR
Description: Weakness measured on a 1-9 scale, 1 being minimal, 9 the worst ever experienced. 0=no symptom reported. For analysis the average severity of weakness for each participant was calculated from daily calls made in weeks 3-4 of each period.
Time Frame: Weeks 3-4 of each period
Population: 44 partipants who experienced weakness in either period 1 or period 2 were included in analysis. All treatment group means are extracted from the mixed effects model. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mexiletine: Particiapnts who experienced weakness on mexiletine capsules 200 mg orally three times daily in either period 1 or period 2.
- Placebo: Particiapnts who experienced weakness on placebo capsules orally three times daily in either period 1 or period 2.
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 44 | 44
units on a scale | 1.96 [1.42 to 2.63] | 3.22 [2.52 to 3.98]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-1.67 to -0.861], Standard Deviation 1.27 — Residual standard deviation

4. Secondary Outcome: Patient Reported Tiredness on the IVR
Description: Tiredness measured on a 1-9 scale, 1 being minimal, 9 the worst ever experienced. 0=no symptom reported. For analysis the average severity of tiredness for each participant was calculated from daily calls made in weeks 3-4 of each period.
Time Frame: Weeks 3-4 of each period
Population: 49 partipants who experienced tiredness in either period 1 or period 2 were included in analysis. All treatment group means are extracted from the mixed effects model. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mexiletine: Particiapnts who experienced tiredness on mexiletine 200 mg capsules orally three times daily in either period 1 or period 2.
- Placebo: Particiapnts who experienced tiredness on placebo capsules orally three times daily in either period 1 or period 2.
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 49 | 49
units on a scale | 2.90 [2.12 to 3.68] | 3.82 [3.03 to 4.53]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald; Mean Difference (Final Values) = -0.918, 95% CI 2-sided [-1.30 to -0.532], Standard Deviation 1.29 — Residual standard deviation

5. Secondary Outcome: Quantitative Measure of Hand Grip Myotonia (Seconds)
Description: Maximum voluntary contractions following forced right hand grip were recorded and the time to relax from 90% to 5% of average maximal force was determined using automated analysis software.
Time Frame: The end of period 1 (week 4) and period 2 (week 9)
Population: All participants with quantitative handgrip myotonia values in either period 1 or period 2 were included in analysis. The treatment-specific group mean is a geometric-like mean using log (t+0.1) 'normalizing' transformation. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: seconds
Groups:
- Mexiletine: Average 90% to 5% hand grip relaxation time for particpants receiving mexiletine 200 mg capsules orally three times daily either in period 1 or period 2
- Placebo: Average 90% to 5% hand grip relaxation time for particpants receiving placebo capsules orally three times daily either in period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 54 | 54
seconds | 0.321 [0.274 to 0.370] | 0.429 [0.365 to 0.517]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; P value indicates significance level of the Wald test associated with mexiletine effect from the linear mixed effects model. All P values were 2-sided and .05 was considered the threshold of statistical significance; Test type: Superiority or Other; p < 0.001, Wald; Mean Difference (Final Values) = -0.109, 95% CI 2-sided [-0.177 to -0.056], Standard Deviation 0.563 — Residual standard deviation

6. Secondary Outcome: Compound Motor Action Potentials After Short Exercise Test
Description: The maximal post-exercise compound muscle action potential (CMAP) after short periods of exercise as a percent of the baseline measurement.
Time Frame: The end of period 1 (week 4) and period 2 (week 9)
Population: All participants with short exercise test values in either period 1 or period 2 were included in analysis. The treatment-specific group mean is taken from the mixed model. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: percentage of baseline CMAP amplitude
Groups:
- Mexiletine: Post exercise CMAP amplitude (as a percent of baseline measurement) for particpants receiving mexiletine capsules 200 mg orally three times daily either in period 1 or period 2
- Placebo: Post exercise CMAP amplitude (as a percento f baseline measurement) for particpants receiving mexiletine capsules orally three times daily either in period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 56 | 56
percentage of baseline CMAP amplitude | 83.1 [77.5 to 88.4] | 78.6 [71.9 to 84.7]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.09, wald; Mean Difference (Final Values) = 4.54, 95% CI 2-sided [-0.680 to 9.75], Standard Deviation 13.1 — Residual standard deviation

7. Secondary Outcome: Graded Myotonia by Needle Electromyography - Right Abductor Digiti Minimi
Description: Measured the amount of myotonia present on needle exam by assigning a number 1-3, with 1 being minimal amount of myotonia on needle stick and 3 being maximal amount of myotonia present on needle stick.
Time Frame: The end of period 1 (week 4) and period 2 (week 9)
Population: All participants with graded needle EMG of the RADM values in either period 1 or period 2 were included in analysis. The treatment-specific group mean is taken from the mixed model. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mexiletine: Graded myotonia in right ADM for particpants receiving mexiletine capsules 200 mg orally three times daily either in period 1 or period 2
- Placebo: Graded myotonia in right ADM for particpants receiving placebo capsules orally three times daily either in period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 56 | 56
units on a scale | 2.05 [1.75 to 2.33] | 2.62 [2.39 to 2.86]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; P value indicates significance level of the Wilcoxon test associated with mexiletine effect from the linear mixed effects model. The Wilcoxon test was substituted because the outcome is not continuous and therefore normality of the residuals is not satisfied. All P values were 2-sided and .05 was considered the threshold of statistical significance; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.568, 95% CI 2-sided [-0.812 to -0.325], Standard Deviation 0.600 — Residual standard deviation

8. Secondary Outcome: Clinical Hand Grip Myotonia Evaluation (Seconds)
Description: The time to open the fist after a forced handgrip as measured on a stopwatch.
Time Frame: The end of period 1 (week 4) and the end of period 2 (week 9)
Population: All participants with clinical handgrip myotonia values in either period 1 or period 2 were included in analysis. The treatment-specific group mean is a geometric-like mean. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: Seconds
Groups:
- Mexiletine: Average time to open the fist after forced hand grip for particpants receiving mexiletine 200 mg capsules orally three times daily either in period 1 or period 2
- Placebo: Average time to open the fist after forced hand grip for particpants receiving placebo capsules orally three times daily either in period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 57 | 57
Seconds | 0.164 [0.0858 to .294] | 0.494 [0.281 to 0.872]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald; Mean Difference (Final Values) = -0.330, 95% CI 2-sided [-0.633 to -0.142], Standard Deviation 1.083 — Residual standard deviation

9. Secondary Outcome: Clinical Eye Closure Myotonia Evaluation (Seconds)
Description: Time to open the eyes after forced eye closure as measured on a stopwatch.
Time Frame: The end of period 1 (week 4) and the end of period 2 (week 9)
Population: All participants with clinical eye closure myotonia values in either period 1 or period 2 were included in analysis. The treatment-specific group mean is a geometric-like mean. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: Seconds
Groups:
- Mexiletine: Average time to open eyes after forced eye closure for particpants receiving mexiletine 200 mg capsules orally three times daily either in period 1 or period 2
- Placebo: Average time to open eyes after forced eye closure for particpants receiving placebo capsules orally three times daily either in period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 57 | 57
Seconds | 0.161 [0.0704 to 0.314] | 0.474 [0.261 to 0.871]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald; Mean Difference (Final Values) = -0.313, 95% CI 2-sided [-0.602 to -0.149], Standard Deviation 0.889 — Residual standard deviation

10. Secondary Outcome: Graded Myotonia by Needle Electromyography - Right Tibialis Anterior
Description: as for outcome 7
Time Frame: The end of period 1 (week 4) and period 2 (week 9)
Population: All participants with graded needle EMG of the RTA values in either period 1 or period 2 were included in analysis. The treatment-specific group mean is taken from the mixed model. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mexiletine: Graded myotonia in right TA for particpants receiving mexiletine capsules 200 mg orally three times daily either in period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 56 | 56
units on a scale | 2.07 [1.73 to 2.37] | 2.54 [2.28 to 2.76]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.464, 95% CI 2-sided [-0.675 to -0.254], Standard Deviation 0.516 — Residual standard deviation

11. Secondary Outcome: Compound Motor Action Potentials After Long Exercise Test
Description: Compound muscle action potential (CMAP) after long periods of exercise as a percentage of baseline.
Time Frame: The end of period 1 (week 4) and period 2 (week 9)
Population: All participants with long exercise test values in either period 1 or period 2 were included in analysis. The treatment-specific group mean is taken from the mixed model. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: percentage of baseline CMAP amplitude
Groups:
- Mexiletine: Post exercise CMAP amplitude (as a percentage of baseline measreument) for participants receiving mexiletine capsules 200 mg orally three times daily either in period 1 or period 2
- Placebo: Post exercise CMAP amplitude ( as a percentage of baseline measurement) for participants receiving placebo capsules orally three times daily either in period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 56 | 56
percentage of baseline CMAP amplitude | 81.8 [76.8 to 87.0] | 80.1 [74.7 to 86.4]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.50, wald; Mean Difference (Final Values) = 1.69, 95% CI 2-sided [-3.34 to 6.73], Standard Deviation 12.6 — Residual standard deviation

12. Secondary Outcome: Individualized Neuromuscular Quality of Life Scale - Summary Score
Description: Quality of life scale for patinets with neuromuscular disorders. The INQoL summary score is a weighted average made up of 5 subdomains (activities, social relationships, independence, emotions, and body image) which document the impact of a disease on a patients' quality of life. Scores range from 0-100, and can be interpreted as the percent of maximal detrimental impact on quality of life. A higher score indicates more detrimental impact.
Time Frame: The end of period 1 (week 4) and period 2 (week 9)
Population: All participants with INQoL summary score values in either period 1 or period 2 were included in analysis. The treatment-specific group mean is taken from the mixed model. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mexiletine: INQoL summary score for participants receiving mexiletine capsules 200 mg orally three times daily either in period 1 or period 2
- Placebo: INQoL summary score for participants receiving placebo capsules orally three times daily either in period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 51 | 51
units on a scale | 14.0 [11.6 to 16.5] | 16.7 [14.0 to 19.4]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, wald; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-4.07 to -1.30], Standard Deviation 3.44 — Residual standard deviation

13. Secondary Outcome: Short Form 36 - Physical Composite Score
Description: The SF-36 is a standard quality of life instrument. The physical composite score represents the the physical burden on quality of life and is a summary of questions related to physical impact of a disease or condition (physical function, role physical, bodily pain, and general health). The score is nomralized to the population and ranges from 0-100, with the US normal value of 50. A lower score represents a greater impact of quality of life.
Time Frame: Particiapnts who experienced weakness on mexiletine in either period 1 or period 2.
Population: All participants with SF-36 physical composite values in either period 1 or period 2 were included in analysis. The treatment-specific group mean is taken from the mixed model. Confidence intervals are bootstrap confidence intervals.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mexiletine: SF-36 physical composite score for participants receiving mexiletine capsules 200 mg orally three times daily either in period 1 or period 2
- Placebo: SF-36 physical composite score for participants receiving placebo capsules orally three times daily either in period 1 or period 2
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 57 | 57
units on a scale | 44.8 [41.9 to 47.4] | 39.2 [35.9 to 41.9]
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, wald; Mean Difference (Final Values) = 5.58, 95% CI 2-sided [3.44 to 7.72], Standard Deviation 5.35 — Residual standard deviation

14. Secondary Outcome: Short Form 36 - Mental Composite Score
Description: The SF-36 is a standard quality of life instrument. The mental composite score represents the the mental burden on quality of life and is a summary of questions related to mental impact of a disease or condition (mental function, role emotional, vitality, and mental health). The score is nomralized to the population and ranges from 0-100, with the US normal value of 50. A lower score represents a greater impact of quality of life.
Time Frame: The end of period 1 (week 4) and period 2 (week 9)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mexiletine - Period 1: SF-36 mental composite for participants receiving mexiletine capsules 200 mg orally three times daily in period 1. Due to an interaction between period and treatment the primary outcome was presented separately for periods 1 and 2.
- Placebo - Period 1: SF-36 mental composite for participants receiving placebo capsules orally three times daily in period 1. Due to an interaction between period and treatment the primary outcome was presented separately for periods 1 and 2.
- Mexiletine - Period 2: SF-36 mental composite for participants receiving mexiletine capsules 200 mg orally three times daily in period 2. Due to an interaction between period and treatment the primary outcome was presented separately for periods 1 and 2.
- Placebo - Period 2: SF-36 mental composite for participants receiving placebo capsules orally three times daily in period 2. Due to an interaction between period and treatment the primary outcome was presented separately for periods 1 and 2.
Arm/Group | Mexiletine - Period 1 | Placebo - Period 1 | Mexiletine - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 28 | 29 | 29 | 25
units on a scale | 47.4 [44.0 to 50.2] | 47.7 [44.2 to 51.3] | 53.1 [50.3 to 55.8] | 42.7 [36.8 to 48.3]
Statistical Analysis 1: Comparison: Mexiletine - Period 1 vs Placebo - Period 1; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.90, Wald; Mean Difference (Final Values) = -0.351, 95% CI 2-sided [-5.87 to 5.17], Standard Deviation 6.50 — Residual standard deviation
Statistical Analysis 2: Comparison: Mexiletine - Period 2 vs Placebo - Period 2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.03, wald; Mean Difference (Final Values) = 10.4, 95% CI 2-sided [0.941 to 20.6], Standard Error of Mean 6.50 — Residual standard deviation

ADVERSE EVENTS:
Time Frame: Data was collected over a 3 year period
Groups:
- Mexiletine Treatment: Adverse events that occurred when patients were taking placebo.
- Placebo Treatment: Adverse events that occurred when patients were taking mexiletine.
Arm/Group | Mexiletine Treatment | Placebo Treatment
Serious Adverse Events (participants affected / at risk) | 1/57 | 0/57
Other Adverse Events (participants affected / at risk) | 24/57 | 11/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mexiletine Treatment (N=57) | Placebo Treatment (N=57)
Drug withdrawal (Psychiatric disorders) | 1/1 (1) | 0/0 (0) — Admitted for withdrawal of narcotics due to pregnancy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexiletine Treatment (N=57) | Placebo Treatment (N=57)
Constitutional (General disorders) | 3 (3) | 0 (0)
Dermatologic/skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 9 (9) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 3 (3)
Lymphatics (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Musculosketetal/soft tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neurologic (Nervous system disorders) | 5 (5) | 1 (1)
Pain (General disorders) | 4 (4) | 0 (0)
Cardiac (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No